CLINICAL TRIAL: NCT01833091
Title: Creating an Artificial Night on Physiological Changes in Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, vajihe sanadgol, principal investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Artificial Night
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-03

CONDITIONS: Physiologic Changes
MeSH Terms: interventions — Light Pollution; Methods

ARMS (2):
- intervention (Experimental): creat light period 12 hours with cover on incubator
  Interventions: Other: artificial night
- control (No Intervention)

INTERVENTIONS:
Other: artificial night — Infants in the intervention group received light cyclic with pattern 12 hours. Light period was from 7 to 19 during which the infants were put in the normal environmental light and dark period was from 19 to 7 during which was the infants' incubator was covered with linen cloth. The vital signsand & arterial oxygen saturation of the infants in the intervention group were controlled before covering the incubator i.e. at 19. Also, the infant's vital signs were again monitored at 7 am.The infant weighed in every day at 7 am during the 10 days of study. Feeding tolerance was daily determined at 8 am, using nasogastric tube or orogastric tube to control residue as well as to review the presence or absence of abdominal distention, vomiting.
  Other Names: intervention
  Arms: intervention

SUMMARY:
Effects of creating an artificial night on physiological changes, weight and feeding tolerance in preterm infants.

Introduction:Nowdays,with medical advances in intensive care increased chance of survival in premature infants.One of the major concerns exposure to high light levels in neonate & subsequent it is increase in metabolism rate.So,this study was conducted to determine the effect of creating an artificial night on physiological changes, weight and feeding tolerance in preterm infants.

Methods: This is a randomized clinical trial dual group study, 38 preterm infants (gestational age of 30-34weeks)due to prematurity hospitalized at Ghaem NICU,were evaluated within 10 days. Infants were divided into two groups of 1200-1700 and 1701-2200g based on the weight and the weight of each group were randomized into artificial night(dark period was from 19 to 7 during incubator was covered with linen cloth & light period was from 7 to 19 removed the cover) and control groups(continuous lighting). Mothers & infants through questionnaires,interviews,observation & document completion, changes in physiologic & weight befor entering the study & then physiologic changes twice a day,weight & feeding tolerance were collected daily.Data were analyzed using spss v.16 software.

ELIGIBILITY:
Inclusion Criteria:

Premature newborn infants with gestational age of 30-34 weeks Birth weight of 1200-2200g Taking care and supervision in the incubator to measure weight and grow up Keeping the axillary temperature in the range of 36-37° C Keeping the heart rate in the range of 100 to 160 beats per minute Breast feeding through a nasogastric tube or gastric orally Healthy infants without congenital anomalies No history of taking specific drugs or alcohol by mother during the pregnancy. Mother's lack of addiction

Exclusion Criteria:

Illness of the infant (affecting with secondary sepsis, seizures; increased or decreased blood pressure, successive apnea, feeding intolerance or feeding stoppage) Starting phototherapy Discharge of the infant earlier than 10 days Parents' lack of consent with the study

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
effect of creating an artificial night on physiological changes, weight and feeding tolerance in preterm infants | 1 years
  physiological changes including:systolic blood pressure & diastolic blood pressure(mm/hg),resoiratory rate(number of minutes),pulse rate(beats per minute), temperature(° C),arterial oxygen saturation(percent),daily weighting & comparing it with the previous days(gram),feeding tolerance(residual volume,vomiting,abdominal distention)

REFERENCES:
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174